CLINICAL TRIAL: NCT03163498
Title: Sleep, Mood and Physical Activity Level in Patients With Hypertension
Brief Title: Evaluation of Sleep Pattern and Mood Profile in Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Professor, Universidade Federal de Goias
Other Study IDs: 1.986.587
Record Dates: First submitted 2017-05-20; First posted 2017-05-23 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Sleep
Keywords: Hypertension; Exercise; Sleep
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACTIVE: Participating in this group will be 30 active hypertension patients who exercise at least 3 times a week for at least 30 minutes
  Interventions: Other: No intervantion. It´s a Cross-Sectional Study
- INACTIVE: Participating in this group will be 30 inactive hypertension patients who do not exercise.
  Interventions: Other: No intervantion. It´s a Cross-Sectional Study

INTERVENTIONS:
Other: No intervantion. It´s a Cross-Sectional Study — No intervential

SUMMARY:
Introduction: Sleep disturbances may contribute to impairments in mood, occupational and intellectual performance, and social relationships, as well as being associated with cardiovascular diseases, such as arterial hypertension. Sedentary lifestyle has often been associated with poor sleep quality and hypertension; regular exercise has been studied as a coadjuvant therapy for hypertension and/or for some sleep disorders. Objective: To compare sleep pattern of active and inactive patients with arterial hypertension, as well as to evaluate complaints of depression and anxiety, and the mood profile. Material and Methods: Polysomnography, Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale will be used to assess the sleep pattern. Depression will be assessed by the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI) anxiety, and mood pattern by the State of Mood Profile (POMS). The level of physical activity will be recorded by the number of steps taken (pedometer). Participating in the study will be 60 hypertension patients (ACTIVE, n=30; INACTIVE, n=30). Hypothesis: Active hypertensive patients better quality of sleep, better mood profile, and fewer complaints of depression and anxiety when compared to physically inactive hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic arterial hypertension, according to the VII Brazilian Guidelines for Hypertension;
* male;
* BMI <30;
* Age between 30 and 60 years;
* Minimum level of education: elementary school

Exclusion Criteria:

* Present pathologies in the musculoskeletal and neurological systems, or incapacitating complaints in these systems;
* Diagnosis of psychiatric disorder;
* Being under medical treatment for insomnia or other psychiatric treatment.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participating in the study will be 60 males hypertension patients (ACTIVE, n=30; INACTIVE, n=30) with age between 30 and 60 years old. All participants should be under antihypertensive drug treatment.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Sleep | 3 months
  Polysomnography, Pittsburgh Sleep Quality Index
Exercise | 3 months
  Normal Physical Activity Level, Pedometer
Mood | 3 months
  Profile of Mood States
Anxiety | 3 months
  Beck Anxiety Inventory
Depression | 3 months
  Beck Depression Inventory
Daytime drowsiness | 3 months
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Passos, PHD, Principal Investigator — World Health Organization
Locations (1):
- Anna Paula Ribeiro Campos, Rio Verde, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Passos GS, Poyares D, Santana MG, Teixeira AA, Lira FS, Youngstedt SD, dos Santos RV, Tufik S, de Mello MT. Exercise improves immune function, antidepressive response, and sleep quality in patients with chronic primary insomnia. Biomed Res Int. 2014;2014:498961. doi: 10.1155/2014/498961. Epub 2014 Sep 21. PMID 25328886
- [Background] Passos GS, Poyares DL, Santana MG, Tufik S, Mello MT. Is exercise an alternative treatment for chronic insomnia? Clinics (Sao Paulo). 2012;67(6):653-60. doi: 10.6061/clinics/2012(06)17. PMID 22760906
- [Result] Passos GS, Santana MG, Poyares D, D'Aurea CV, Teixeira AA, Tufik S, de Mello MT. Chronotype and anxiety are associated in patients with chronic primary insomnia. Braz J Psychiatry. 2017 Apr-Jun;39(2):183-186. doi: 10.1590/1516-4446-2016-2007. Epub 2017 Jan 9. PMID 28076650